CLINICAL TRIAL: NCT06358430
Title: Phase 1 Dose Escalation and Expansion Study of TROP2 CAR Engineered IL-15- Transduced Cord Blood-derived NK Cells in Combination With Cetuximab in Patient With Colorectal Cancer (CRC) With Minimal Residual Disease (MRD)
Brief Title: Dose Escalation and Expansion Study of TROP2 CAR Engineered IL-15- Transduced Cord Blood-derived NK Cells in Combination With Cetuximab in Patient With Colorectal Cancer (CRC) With Minimal Residual Disease (MRD)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bellicum Pharmaceuticals, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-1017; NCI-2024-03107 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer; Minimal Residual Disease
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm, Residual | interventions — fludarabine phosphate; fludarabine; Cyclophosphamide; Cetuximab; AP 1903 reagent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation + Dose Expansion (Experimental): Up to 5 dose levels of TROP2-CAR-NK cells will be tested in the Dose Escalation phase. Up to 12 participants maximum will be enrolled at any dose level, in groups of 3 participants at a time. The first group of participants will receive the lowest dose level.
  Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the recommended dose of TROP2-CAR-NK cells is found. When that dose level is confirmed, the final group of 12 participants will be enrolled at that dose level.
  Interventions: Drug: Fludarabine Phosphate; Drug: Cyclophosphamide; Drug: Cetuximab; Drug: TROP2-CAR-NK Cells; Drug: Rimiducid (AP1903); Procedure: Lymphodepleting Chemotherapy

INTERVENTIONS:
Drug: Fludarabine Phosphate — Given by IV
  Other Names: Fludarabine; Fludara®
Drug: Cyclophosphamide — Given by IV
  Other Names: Cytoxan®; Neosar®
Drug: Cetuximab — Given by IV
  Other Names: C225; Erbitux™; IMC-C225; MOAB C225
Drug: TROP2-CAR-NK Cells — Given by IV
Drug: Rimiducid (AP1903) — Given by IV
Procedure: Lymphodepleting Chemotherapy — Given by Chemotherapy

SUMMARY:
To find the highest and/or recommended dose of TROP2-CAR-NK cells combined with cetuximab in participants with MRD CRC.

DETAILED DESCRIPTION:
Primary Objective:

1. To determine the safety, tolerability, maximum tolerated dose (MTD), and recommended Phase 2 dose (RP2D) of TROP2-CAR-NK cells combined with cetuximab in patients with MRD CRC.
2. To evaluate circulating tumor DNA (ctDNA) clearance (undetectable) at 3 months

Secondary Objectives:

1. Determine progression-free survival.
2. To quantify the persistence of infused allogeneic donor TROP2-CAR-NK cells in the peripheral blood of the recipient.
3. To evaluate blood- and tissue-based biomarkers at baseline associated with response and resistance to TROP2-CAR-NK cell infusion in combination with cetuximab.

Exploratory Objectives:

1. To profile and assess dynamic immune changes in the tumor microenvironment.
2. Quantify the average circulating ctDNA change from TROP2-CAR-NK infusion to progression or initiation of a new cancer therapy and association with PFS.
3. To evaluate patient-reported quality of life (QoL).

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be 18 years or older.
2. Participants must be willing and able to provide informed consent.
3. Willing and able to comply with clinical trial instructions and requirements. Individuals lacking the ability, based on reasonable medical judgment, to understand and appreciate the nature and consequences of participation in this study will not be eligible for participation.
4. In both the dose escalation and dose expansion cohorts, participants must have documented colorectal cancer (CRC) with MRD following complete disease resection followed by standard-of-care adjuvant treatment. MRD is defined as NO evidence of radiological disease (including patients with undefinable lesion with max diameter <1 cm or with a short axis < 1cm for lymph nodes) and presence of circulating ctDNA in the bloodstream.
5. Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (Appendix 3).
6. Life expectancy > 3 months.
7. A female patient is eligible to participate if at least one of the following conditions applies:

   * Not a woman of childbearing potential (WOCBP) as defined in Appendix 4 OR
   * A WOCBP who agrees to follow the contraceptive guidelines in Appendix 4 during the study treatment period and for 6 months post TROP2-CAR-NK cell infusion.
8. Female participants who become pregnant or suspect pregnancy must immediately notify their doctor. Females' participants who become pregnant will be taken off study.
9. Male participants must agree to follow the contraceptive guidelines in Appendix 4 during the study treatment period and for 6 months post TROP2-CAR-NK cell infusion. Male participants who father a child or suspect that they have fathered a child must immediately notify their doctor.
10. WOCBP must have a negative urine pregnancy test within 72 hours prior to the start of lymphodepleting chemotherapy. If a WOCBP has a urine pregnancy test that cannot be confirmed as negative, a serum (beta-human chorionic gonadotropin [â-hCG]) pregnancy test will be required.
11. Participants must have adequate organ function as defined below (Table 1) within 10 days prior to the start of lymphodepleting chemotherapy:

    Table 1. Adequate Organ Function Laboratory Values Systemic Function Test Laboratory Value Hematologic ANC = ≥1500/ƒÊL Platelets = ≥100,000/ƒÊL Hemoglobin = ≥9.0 g/dLa Renal CrCl by Cockcroft-Gault formula = ≥45 mL/min for patients with creatinine >1.5 x ULNb Hepatic Total bilirubin = ≤1.5 x ULN OR direct bilirubin ≤ULN for patients with total bilirubin levels >1.5 x ULN AST and ALT = ≤2.5 x ULN (≤5 x ULN for patients with history of resected liver metastases) Coagulation PT/INR aPT = ≤1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range
12. Left ventricular ejection fraction >50%. Of note, those patients with risk factors and/or with LVEF <55% additional testing may need to be performed as per institutional guidelines and/or PI guidance.
13. Adequate respiratory reserve defined as dyspnea Grade 0 or 1 and saturated oxygen >92% in room air.
14. Willing to undergo mandatory blood collections and biopsies as required by the study.
15. Willing to stay within a 2-hour drive (approximately 100-mile radius) of the study site during the first 4 weeks after the TROP2-NK cell infusion.

Exclusion Criteria:

1. Participants with known active disease by RECIST v1.1.
2. Pregnant, breastfeeding, or expecting to conceive within the projected duration of the study, starting with the screening visit through 6 months post TROP2-CAR-NK cell infusion.
3. Has received systemic anticancer therapy within 2 weeks or 3 half-lives, whichever is shorter, prior to the start of lymphodepleting chemotherapy. For patients treated with monoclonal antibodies, at least 3 weeks must have elapsed prior to the start of lymphodepleting chemotherapy. Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 3 weeks after the last dose of the previous investigational agent.
4. Participants must have recovered from all AEs due to previous therapies to . Grade 1 or baseline. Participants with ≤ Grade 2 neuropathy, alopecia, or other non-relevant AEs may be deemed eligible at the discretion of the principal investigator (PI). If a participants received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to the start of lymphodepleting chemotherapy.
5. Has received prior radiotherapy within 2 weeks of the start of lymphodepleting chemotherapy. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis or colitis.
6. Has received a live vaccine within 6 weeks prior to TROP2-CAR-NK infusion and for at least 24 months post infusion. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette. Guerin, and typhoid vaccine. Seasonal influenza and COVID-19 vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMistR) are live attenuated vaccines and are not allowed.
7. Prior genetically modified T or NK cell therapy.
8. Has diagnosis of immunodeficiency or receiving chronic systemic steroid therapy (in doses exceeding 10 mg daily of prednisone equivalent).
9. History of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years. The time requirement does not apply to patients who underwent successful definitive resection of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, in situ cervical cancer, or other in situ cancers.
10. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is allowed.
11. History of interstitial lung disease (ILD) that required steroids or has current pneumonitis/ILD.
12. Active infection requiring systemic therapy.
13. Known human immunodeficiency virus (HIV) infection.
14. Known active or chronic hepatitis B or hepatitis C virus infection.
15. Known history of active tuberculosis (Mycobacterium Tuberculosis).
16. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participants to participate, in the opinion of the treating investigator.
17. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
18. Has had an allogenic tissue/solid organ transplant.
19. Clinically significant cardiovascular disease within 12 months prior to the start of lymphodepleting chemotherapy, including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebrovascular event, or cardiac arrhythmia associated with hemodynamic instability. NOTE: medically controlled arrhythmia would be permitted if meet criteria per Appendix X.
20. Prolongation of corrected QT interval using Fridericia's formula to >480 milliseconds, unless cleared after cardiology evaluation.
21. Participant with bleeding or thrombotic disorders or at risk for severe hemorrhage. Participants with known deep vein thrombosis/pulmonary embolism who are on appropriate anti-coagulation treatment are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2029-01-18 (Estimated); Study Completion 2029-01-18 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Maria Pia Morelli, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org